CLINICAL TRIAL: NCT07149337
Title: Assessing Human Phosphate Tolerance and Its Dependency on Age and Sex
Brief Title: Assessing How the Body Responds to Increased Phosphate Intake, and How This Response Depends on Age and Sex.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-02538
Record Dates: First submitted 2025-08-22; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Aging; Kidney Disease; Mineral Metabolism
Keywords: Phosphate homeostasis and aging; Oral phosphate challenge
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral phosphate load (Experimental): Participants will eat a standard phosphate dinner. The next morning, after consuming a standard phosphate breakfast, they will ingest a phosphate load (558 mg phosphorus) and provide blood and urine samples for nine hours.
  Interventions: Other: Oral phosphate load

INTERVENTIONS:
Other: Oral phosphate load — Participants ingest an oral phosphate load containing 558 mg of phosphorus once.

SUMMARY:
Kidney function declines with age and this could affect phosphate balance after an acute phosphate load (increased phosphate intake). In daily life, we regularly experience acute phosphate loads through our diet.

The aim of this clinical study is to determine whether the body's response to increased phosphate intake changes with age and whether there are sex differences in this response.

DETAILED DESCRIPTION:
Forty subjects (males and females aged 18-25 or 63-70) will ingest an oral phosphate load, after which their body's response will be assessed by collecting blood and urine samples over a period of ten hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 18-25 and 63-70 years old
* 18.5 ≥ BMI < 26 kg/m2
* 0.84 ≥ phosphate in plasma ≤ 1.45 mM
* 2.20 ≥ calcium in plasma ≤ 2.50 mM
* 15 ≥ PTH in plasma ≤ 65 pg/ml
* eGFR ≥ 60 ml/min/1-73 m2
* 90 ≥ Systolic blood pressure ≤ 140 mmHg
* 60 ≥ Diastolic blood pressure ≤ 85 mmHg
* No hematuria and no acute urinary tract infection
* Ability and willingness to participate in the study
* Voluntary signed inform consent

Exclusion Criteria:

* Diabetes mellitus
* Pregnancy
* History of kidney stones
* History of parathyroidectomy
* History of anorexia nervosa
* History of bulimia
* History of solid organ transplantation.
* Nephrolithiasis
* Sarcoidosis
* Chronic pancreatitis
* Chronic diarrhea
* Chronic liver disease
* Complete distal renal acidosis (dRTA)
* Cystinuria
* Hypo- or hyperaldosteronism
* Hyper- or hypotension
* Hypernatremia
* Gastrointestinal disorders
* Known hypersensitivity reactions to azoic dyes, acetylsalicylic acid, as well as antirheumatic drugs and painkillers (prostaglandin synthesis inhibitors).

Intake of vitamin D and calcium supplements, phosphate, bisphosphonates, cinacalcet, denusomab, teriparatide, systemic glucocorticoids or mineralcorticoids, antiepileptics, carboanydrase inhibitors or diuretics

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Phosphate in plasma | The primary outcome will be measured 5 hours after the first blood collection on the day of the study and 4 hours after ingesting the oral phosphate load.
  Phosphate in plasma 4 hours after the oral phosphate load shows age differences